CLINICAL TRIAL: NCT04695886
Title: Evaluation of the Effectiveness and Cost-effectiveness of a Community-delivered Integrated Malaria Elimination (CIME) Model in Myanmar: An Open Stepped-wedge Cluster-randomised Controlled Trial
Brief Title: Effectiveness of a Community-delivered Integrated Malaria Elimination (CIME) Model in Myanmar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: National Malaria Control Program, Myanmar (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 241/20_CIME_Malaria
Record Dates: First submitted 2020-12-19; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Malaria
Keywords: Community-delivered; Intervention; elimination; falciparum; vivax; routine testing; Stepped-wedge
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized control trial (one-way crossover)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIME intervention (Experimental): Community-delivered Integrated Malaria Elimination (CIME). The CIME intervention model integrates interventions for malaria, dengue, tuberculosis, childhood diarrhoea and RDT-negative fever.
  Interventions: Other: Community-delivered Integrated Malaria Elimination (CIME) intervention model
- ICMV standard of care (No Intervention): Integrated Community Malaria Volunteer (ICMV) model - this is the current standard of care. This model involves malaria volunteers undertaking additional screening and referral services for a range of other diseases including: dengue, lymphatic filariasis, tuberculosis, HIV/AIDS and leprosy.

INTERVENTIONS:
Other: Community-delivered Integrated Malaria Elimination (CIME) intervention model — Malaria: Malaria Diagnosis using RDT, treatment, referral and reporting; Prevention interventions (Behavioral Change Communication, net and repellent distribution); assisting in case and foci investigation and larval source management.
  Dengue: Assisting in dengue prevention; Referral of cases. Tuberculosis (TB): Detection and referral of suspected cases; Contact tracing; Directly observed treatment, short-course (DOTS) providers; defaulter tracing; follow-up sputum examinations; assisting in TB health education talks and active case detection activities.
  Childhood diarrhea: Prevention; Health education and Water, sanitation and hygiene (WASH) promotion; Diagnosis and dehydration assessment; Treatment and referral; Rehydration therapy using Oral Rehydration Solution (ORS) and oral Zinc tablet; assisted referral.
  RDT-negative fever: Prevention and health education; Symptomatic treatment with antipyretics and immediate assisted referral.
  Arms: CIME intervention

SUMMARY:
In Myanmar, community health workers, known as malaria volunteers, have played a key role in reducing the malaria burden in the malaria control phase, providing essential malaria services in rural areas where the coverage of formal health services is limited. However, the community-delivered models that have worked well for malaria control may not work well for malaria elimination. In parallel with switching from interventions for malaria control to those for elimination, the motivation and social importance of malaria volunteers has declined along with the decline of the malaria burden. To sustain volunteer motivation, the social importance and effectiveness in the malaria elimination program, the Community-delivered Integrated Malaria Elimination model for Myanmar (CIME model) was developed based on global evidence and qualitative consultations with community members, leaders, volunteers and health stakeholders in Myanmar. This study will assess the level of effectiveness of the CIME model in increasing malaria testing by its application in an open cluster-randomised controlled stepped-wedge trial.

DETAILED DESCRIPTION:
The CIME model integrates interventions for malaria, dengue, tuberculosis, childhood diarrhoea and Rapid Diagnostic Test (RDT)-negative fever. It will involve the recruitment and training of a volunteer to implement the CIME model in each village.

The primary outcome of the trial is blood examination rate as determined by number of RDTs for malaria performed per week per village. 140 villages in 8 townships across Ayeyarwaddy, Bago and Yangon Regions and Kayah State in Myanmar will be sampled at random with probability proportional to size. Study populations include villages with ICMVs who will be re-trained as CIME volunteers (intervention phase) and the community members in the service catchment areas of those volunteers. An open stepped-wedge cluster-randomised controlled trial, randomized at the volunteer level (i.e. the volunteer and the village / workplaces they service), will be conducted over 6-months to evaluate the effectiveness and cost-effectiveness of the CIME model intervention. The stepped-wedge design will comprises 24 weekly measurements of the number of malaria blood examinations performed by each village, with villages grouped into 10 blocks of 14 villages and transitioned from control to intervention phases at bi-weekly intervals following a universal two-week control period. Differences in the per weekly rate of blood examination (primary outcome), will be estimated across intervention and control phases using a generalised linear (e.g. Poisson or negative-binomial link functions) mixed modelling analytical approach with maximum likelihood estimation.

ELIGIBILITY:
Inclusion Criteria:

* Villages in Ayeyarwaddy, Bago and Yangon Regions and Kayah State townships in Myanmar with National Malaria Control Program (NMCP) trained Integrated Community Malaria Volunteers (ICMVs).

Exclusion Criteria:

* Townships

A township will be excluded from the study if:

1. The township does not have an NMCP provided ICMV network
2. The township has ongoing armed conflict
3. The township does not have Vector-Borne Diseases Control (VBDC) staff or malaria focal person
4. The location of the township is not geographically or politically feasible for staff from the State/Regional capital city to conduct regular supervision visits

Villages

After selection of 8 townships (2 townships from each state/region), villages in the townships will be screened against the exclusion criteria. A village will be excluded from the study if:

1. The village is too remote and unable to execute the CIME model completely,
2. The village has a government public health facility,
3. The village has no mobile network coverage
4. The village is in the ongoing armed conflict zone , or
5. The village has an ICMV program operated by any organizations other than NMCP
6. The village has an Annual Parasite Index (API) >=5

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6440 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Blood examination rate | Assessed weekly, longitudinally over 6-months
  Change in blood examination rate as determined by the number of rapid diagnostic tests (RDTs) for malaria performed per week per village

SECONDARY OUTCOMES:
Plasmodium spp. infection detected by RDT | Assessed weekly, longitudinally over 6-months.
  Change in the number of Plasmodium spp. infections detected by RDT per week per village
Plasmodium spp. infections reported with 24 hours | Assessed weekly, longitudinally over 6-months.
  Change in the number and percentage of Plasmodium spp. infections reported within 24 hours of RDT per village
Plasmodium spp. infection detected by PCR | Assessed weekly, longitudinally over 6-months.
  Change in the number of Plasmodium spp. infections detected by polymerase chain reaction (PCR) (from RDT cassette) per week
Larval source management | Assessed weekly, longitudinally over 6-months.
  Change in the number of larval sources managed by the volunteer per week
Dengue cases | Assessed weekly, longitudinally over 6-months.
  Change in the number of suspected Dengue cases referred to the nearby clinic per week
Tuberculosis (TB) cases | Assessed weekly, longitudinally over 6-months
  Change in the number of suspected tuberculosis cases referred for diagnosis to national tuberculosis program per week
TB DOTS | 6-month
  Number of TB patients monitored by volunteer for DOTS over the whole study period
Diarrheal cases diagnosed, treated and referred | Assessed weekly, longitudinally over 6-months
  Change in the number of diarrheal cases diagnosed, treated with ORS and zinc tablets and referred per week
RDT-negative fever cases | Assessed weekly, longitudinally over 6-months
  Change in the number of RDT-negative fever cases referred per week
Malaria treatment according to national policy | Assessed weekly, longitudinally over 6-months
  Change in the proportion of patients with confirmed malaria who received first-line antimalarial treatment according to national policy
Data accuracy and completeness in reporting of malaria cases | Assessed weekly, longitudinally over 6-months
  Change in the number of accurately reported and complete malaria case records according the national malaria case-based reporting format
Malaria drug resistance-associated mutations | Assessed weekly, longitudinally over 6-months
  Change in the proportion of Kelch13 and other resistance mutations detected by PCR from RDT cassettes
Seroprevalence of malaria-associated antibodies | Assessed weekly, longitudinally over 6-months
  Change in the seroprevalence of anti-malarial antibodies detected by enzyme-linked immunosorbent assay (ELISA) from RDT cassette
Levels of malaria-associated antibodies | Assessed weekly, longitudinally over 6-months
  Change in the levels of anti-malarial antibodies detected by enzyme-linked immunosorbent assay (ELISA) from RDT cassette
Acceptability of the CIME model by villagers | 6-month
  Acceptability of the CIME model by villagers assessed by an investigator-developed questionnaire including component constructs such as affective attitude, burden, perceived effectiveness and self-efficacy.
Acceptability of the CIME model by CIME volunteers | 6-month
  Acceptability of the CIME model by CIME volunteers assessed by an investigator-developed questionnaire including component constructs such as affective attitude, burden, perceived effectiveness and self-efficacy.
Acceptability of the CIME model by stakeholders | 6-month
  Acceptability of the CIME model by stakeholders assessed by focus group discussions.
Cost-effectiveness of the CIME model | 6-month
  Cost-effectiveness of the CIME model compared to ICMV model (Cost per unit detection, treatment and notification of a malaria case)

CONTACTS AND LOCATIONS:
Overall Officials: Freya Fowkes, DPhil, Principal Investigator — Burnet Institute; Win Han Oo, PhD, Principal Investigator — Burnet Institute

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available after publication from the data custodian(s) to applicants who provide a sound proposal to The Ethics Review Committee on Medical Research Involving Human Subjects, Department of Medical Research, Myanmar Ministry of Health and Sports (No. 5 Ziwaka Road, Dagon PO Yangon, Myanmar; (+95) 01 375447 extension 118; ercdmr2015@gmail.com) contingent of their approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Supporting information will be published in peer-reviewed journals within 2 years of study completion.
Access Criteria: Supporting information can be requested from study investigators

REFERENCES:
- [Derived] Win Han Oo, Htike W, May Chan Oo, Pwint Phyu Phyu, Kyawt Mon Win, Nay Yi Yi Linn, Tun Min, Ei Phyu Htwe, Aung Khine Zaw, Kaung Myat Thu, Galau NH, Cutts JC, Simpson JA, Scott N, O'Flaherty K, Agius PA, Fowkes FJI. Effectiveness of an expanded role for community health workers on malaria blood examination rates in malaria elimination settings in Myanmar: an open stepped-wedge, cluster-randomised controlled trial. Lancet Reg Health Southeast Asia. 2024 Oct 17;31:100499. doi: 10.1016/j.lansea.2024.100499. eCollection 2024 Dec. PMID 39492851
- [Derived] Oo WH, Thi A, Htike W, Agius PA, Cutts JC, Win KM, Yi Linn NY, Than WP, Hkawng GN, Thu KM, Oo MC, O'Flaherty K, Kearney E, Scott N, Phyu PP, Htet AT, Myint O, Lwin Yee L, Thant ZP, Mon A, Htike S, Hnin TP, Fowkes FJI. Evaluation of the effectiveness and cost effectiveness of a Community-delivered Integrated Malaria Elimination (CIME) model in Myanmar: protocol for an open stepped-wedge cluster-randomised controlled trial. BMJ Open. 2021 Aug 13;11(8):e050400. doi: 10.1136/bmjopen-2021-050400. PMID 34389579